CLINICAL TRIAL: NCT05413902
Title: Efficiency of Multi-Modal Anesthesia (MMA) Protocol in Pain Control and Analgesia in Patients Undergoing Posterior Lumbar Spinal Fusion Surgery
Brief Title: Multi-Modal Anesthesia Protocol in Pain Management of Patients Undergoing Posterior Lumbar Spinal Fusion Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A9630120
Record Dates: First submitted 2022-05-05; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Pain Management; Posterior Spinal Fusion
MeSH Terms: conditions — Agnosia | interventions — Ketorolac Tromethamine; Morphine; Narcotics; Analgesics, Opioid; Orphenadrine; Gabapentin; Acetaminophen; Bupivacaine; Epinephrine; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MMA Protocol Group (Experimental): Preoperative Medications
  1. Orphenadrine 100mg PO once preop
  2. Gabapentin 800mg PO once preop
  3. Toradol 60mg IV once preop
  4. Acetaminophen 1,000mg PO once preop
  Intraoperative Paraspinal Infusion
  1. Bupivacaine 30cc
  2. Epinephrine 1cc
  3. Xylocaine-MPF Intramuscular Inj 0.5% (30cc of Saline Solution)
  Postoperative Medications
  1. Orphenadrine 100mg PO BID
  2. Gabapentin 300mg PO Q6
  3. Toradol 30mg IV Q6hrs*
  4. Methylprednisolone 125mg Q8hrs
  Interventions: Drug: Toradol; Drug: Orphenadrine; Drug: Gabapentin; Drug: Acetaminophen; Drug: Bupivacaine; Drug: Epinephrine; Drug: Xylocaine Injectable Solution; Drug: Methylprednisolone
- Control (opioids) Group (Active Comparator): Postoperative Medication
  1-Morphine 4mg Q4hrs
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Toradol — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Morphine — Provide the standard postoperative morphine dose for pain management as part of the traditional opioid-based pain management regime.
  Other Names: Narcotics; Opioids
  Arms: Control (opioids) Group
Drug: Orphenadrine — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Gabapentin — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Acetaminophen — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Bupivacaine — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Epinephrine — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Xylocaine Injectable Solution — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group
Drug: Methylprednisolone — Provide this drug as part of a multimodal pharmacologic regimen for pain management including multiple drugs mentioned in the group description.
  Other Names: Multimodal Analgesia Protocol
  Arms: MMA Protocol Group

SUMMARY:
This study consisted of a randomized controlled trial designed to evaluate a Multimodal Analgesia (MMA) Protocol on patients undergoing Posterior Spinal Fusion. The purpose is to describe the narcotic requirements and usage during the perioperative period of posterior spinal fusion and instrumentation surgery with the implementation of multimodal anesthesia protocol. The study will consist of two parallel arms, with Group 1 receiving our MMA protocol and Group 2 receiving a traditional opioid-based regime. The primary outcome of this study will be the reported Visual Analog Scale (VAS) for pain at 12, 24, and 48 hours after surgery. We considered that our findings could contribute to the fight against the opioid crisis proving alternatives to opioids as feasible alternatives for pain management even in significant surgery, as is posterior spinal fusion with instrumentation.

DETAILED DESCRIPTION:
After seeking Institutional Review Board (IRB) approval, a randomized clinical trial study will be conducted with a diagnosis of Lumbar stenosis between levels of L1-S1 who underwent operative posterior spinal fusion and instrumentation (PSF) and were admitted to Hospital Universitario de Adultos, San Juan, PR. A sample size of n=50 is considered for each study arm. Three surgeons with Spine orthopedic surgery fellowship will perform all the surgical procedures. Inclusion criteria for eligible patients are lumbar stenosis with levels between L1-S1, no prior surgical treatment of spinal deformity, 30 - 85-years of age, and atraumatic pathology. The patients were considered participants after providing written informed consent. Patients were excluded if they were younger than 30 years old or older than 85 years and had a prior history of chronic opioid abuse, corrective surgery, or traumatic pathology. Patients were divided into two randomly selected groups. A random numerator generator has chosen patients' analgesic protocol, creating two groups in an aleatory manner. Group 1 received a Multimodal Analgesia (MMA) Protocol. Group 2 experienced a traditional analgesia protocol (Narcotics/Opioids). As part of the preoperative care for all patients undergoing PSF, lab work includes complete blood count, complete metabolic panel, and coagulation panel. In addition, all patients were assessed by internal medicine for clearance before surgery. Group 1 received multimodal analgesia, including Toradol 60mg IV, Acetaminophen 1,000mg PO, Orphenadrine 100mg PO, and Gabapentin 800 mg PO prior to surgery. Group 2 will not be given oral analgesia preoperatively. As part of the intraoperative care, group 1 was given: Bupivacaine 30cc, Epinephrine 1c,c, and MPF Intramuscular Inj 0.5% (30cc of Saline Solution) in paraspinal and adjacent areas before surgical incision at the time of timeout. Both study arms received routine postoperative care and were followed daily while admitted to the hospital. Patients in group 1 were treated with a postoperative pain management protocol including Gabapentin 300mg PO Q6hrs, Toradol 30mg IV Q6hrs, Methylprednisolone 125mg Q8hrs, and orphenadrine 100mg PO twice daily. Group 2 received a traditional opioid-based pain management approach with Morphine 4mg Q4hrs. Patients were asked for daily pain levels using 1-10, and IV morphine use as needed will be measured daily. Data Collection will occur intra-hospital during the perioperative period. The study variables retrieved included sociodemographic Information, surgery Duration, surgical approach, levels of instrumentation, type of instrumentation, Surgery blood loss, Complications, Discharge Time, Length of Stay, Comorbidities, and Visual Analog Scale (VAS) for pain score preoperative and postoperative at 12, 24, and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* lumbar stenosis affecting L1-S1
* Requiring Posterior Spinal Fusion Surgery
* Age 30-85 years

Exclusion Criteria:

* younger than 30 years old or older than 85 years
* Chronic Renal Disease
* Hypersensitivity to any medication
* history of chronic opioid abuse.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale reported pain score | At 12 hours, at 24 hours and at 48 hours
  The numeric rating scale is an 11-point scale scored from 0-10 to describe the intensity of pain. Patients verbally select the numeric value that is more consistent with the pain experienced. The value 0 consist of no pain and 10 consist the worst pain experienced in life. Therefore, the higher the value the worst the pain is considered.

SECONDARY OUTCOMES:
Number of Days in Hospital | At discharge, at day 3 on average.
  The number of days in hospital represents the duration of postoperative hospital care from the surgery to discharge.
Rate of Surgical Complications | At discharge, at day 3 on average
  The rate of surgical complications will represent any situation that deviates from the adequate/optimal postoperative history or care until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: José Montañez, MD, Principal Investigator — Department of Orthopaedic Surgery, University of Puerto Rico, Medical Sciences Campus, San Juan, PR
Locations (1):
- Puerto Rico Medical Center - University District Hospital, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. However, data could be shared upon individual researchers' reasonable request.

REFERENCES:
- [Derived] Ramirez-Gonzalez M, Torres-Lugo NJ, Deliz-Jimenez D, Echegaray-Casalduc G, Ramirez N, Colon-Rodriguez E, Carro-Rivera J, De La Cruz A, Claudio-Roman Y, Massanet-Volrath J, Escobar-Medina E, Montanez-Huertas J. Efficacy of an Opioid-Sparing Perioperative Multimodal Analgesia Protocol on Posterior Lumbar Fusion in a Hispanic Population: A Randomized Controlled Trial. J Am Acad Orthop Surg. 2023 Sep 1;31(17):931-937. doi: 10.5435/JAAOS-D-22-00878. Epub 2023 May 15. PMID 37192425